CLINICAL TRIAL: NCT01092676
Title: Regular vs Intermittent Dose Ibuprofen for the Treatment of Ankle Sprains in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-08-502; REB 15517 (Other: Research Ethics Board Number)
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Ibuprofen; Ankle Injuries
Keywords: Pediatrics; Emergency
MeSH Terms: conditions — Ankle Injuries; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Ibuprofen Dosing (Active Comparator): Regular Ibuprofen Dosing throughout 4 days of study
  Interventions: Drug: Ibuprofen Regular Dosing
- PRN Ibuprofen dosing (Active Comparator): As needed Ibuprofen dosing
  Interventions: Drug: PRN dosing Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen Regular Dosing — Regular dosing
  Arms: Regular Ibuprofen Dosing
Drug: PRN dosing Ibuprofen — PRN dosing Ibupofen
  Arms: PRN Ibuprofen dosing

SUMMARY:
Ankle sprains are common in children, and optimal pain management has not been determined.

We hypothesize that children age 7-17 years of age with acute ankle sprain randomized to receive regular dose ibuprofen will show a greater improvement in degree of pain,disability,swelling and tenderness four days following injury as compared to children who take ibuprofen only intermittently for pain relief during the same time period.

DETAILED DESCRIPTION:
Acute ankle sprains are one of the most common musculoskeletal injuries in children and adolescents seeking medical attention. There are an estimated 2 million ankle injuries a year and they represent 20 percent of all sports injuries. Data from the National Hospital Ambulatory Medical Care Survey in 2000 showed approximately 1.375 million visits to emergency departments (ED) in the US due to ankle sprains. This represented about 1.3% of all ED visits. The majority of these injuries occur in young athletes. One epidemiological study showed the prevalence of ankle sprains to be 73% in athletes.

The majority of ankle injuries do not involve bony fractures, rather they involve the soft tissue structures of the ankle joint. An ankle sprain is a stretching, partial or complete tear of the ligaments of the ankle. The most common type of ankle sprain is a lateral sprain, usually caused by an inversion injury. Ankle sprains can be classified as a grade I to III, depending on the severity of the injury. A grade I injury is a slight stretching of the ligament; whereas, a grade III sprain is a complete tear of the ligament.

Treatment of ankle sprains is aimed at decreasing the pain and swelling and protecting the ankle ligaments from further injury. The most commonly used acute management strategy includes the RICE (Rest, Ice, Compression, Elevation) protocol. The pharmacologic treatment of ankle sprains however, remains somewhat unclear. Analgesia with acetaminophen was historically the treatment of choice. However, with the development of over the counter NSAID (non-steroidal anti-inflammatory drug) agents, these have become increasingly popular for the treatment of ankle sprains. NSAIDS are a heterogeneous group of drugs that have analgesic, anti-pyretic, and anti-inflammatory effects. They have been used extensively in both adults and children, with ibuprofen being the most commonly used NSAID in North America. The theoretical advantage of the anti-inflammatory action, in addition to the excellent safety profile in children, has made ibuprofen the treatment of choice for musculoskeletal pain in this population.

Controlled trials in adults of various NSAIDS in ankle sprains have shown mixed results. Although they have shown a beneficial effect compared to placebo, they have not consistently shown a benefit over other analgesic choices. Nonetheless, The American Academy of Orthopedic Surgeons recommends that NSAIDs be used to control pain and inflammation in the treatment of acute ankle sprains.

There is very little evidence for the pharmacologic treatment of ankle sprains in children. A study completed at our centre involving 80 patients with acute ankle sprains showed no beneficial effect of naproxyn over acetaminophen in the treatment of pain. However, a study from Ottawa looking at pain relief in all types of musculoskeletal injury, showed a benefit of ibuprofen over both acetaminophen and codeine for pain control. Despite the scant evidence of the benefit of NSAIDS in pediatric ankle sprains, the American Academy of Pediatrics suggests that NSAIDS "can help reduce swelling and pain" in the treatment of ankle sprains.

There currently are no guidelines recommending a dosing schedule of ibuprofen for acute ankle sprains in children. Whether regularly dosed ibuprofen is beneficial versus as-needed dosing of NSAIDs, remains unclear. Interestingly, an unpublished informal survey of the pediatric emergency physicians at the Children's Hospital of Western Ontario, revealed universal recommendations of RICE therapy and the use of ibuprofen for the treatment of ankle sprains. However, the recommendations for ibuprofen dosing varied widely from as-needed to regular dosing.

The purpose of this study is to examine if regular dosed ibuprofen has an advantage over as-needed dosed ibuprofen in the treatment of acute ankle sprains in children.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-17 years who have suffered an isolated ankle sprain within the last 24 hours
* Able to return for follow-up with research assistant in 4 days time

Exclusion Criteria:

* Preexisting Metabolic bone disease
* Bilateral ankle sprains
* Fractured ankle as demonstrated on X-ray
* Suspected Salter 1 fracture or syndesmosis injury
* Other traumatic injuries
* History of Gastric ulcers or renal disease
* Known or suspected allergy/sensitivity to ibuprofen
* Previous ankle sprain of affected ankle within last 6 months

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrick Lim, MD,FRCPC,FAAP, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regular Ibuprofen Dosing | PRN Ibuprofen Dosing
Started | 50 | 49
Completed | 50 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular Ibuprofen Dosing | PRN Ibuprofen Dosing | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 49 | 99
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Pain on Weight Bearing From Baseline
Description: Change in Pain Scale 0-10 Visual Analog Scale with 0 being no pain and 10 being unbearable pain. Outcome is measured in mm as measured from 0 to where the participant places indicated their pain to be on the scale.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Regular Ibuprofen Dosing | PRN Ibuprofen Dosing
Number analyzed (Participants) | 50 | 49
mm | 6.96 (2.26) | 6.70 (2.17)

2. Primary Outcome: Change in Visual Analog Scale (VAS) for Disability
Description: 0-10 Visual Analog Scale with 0 being no disability and 10 being severe disability. Patients are asked to place a line on the VAS to where they believe their disability to be. The final outcome is then measured in mm from 0 to the line placed by the patient.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Regular Ibuprofen Dosing | PRN Ibuprofen Dosing
Number analyzed (Participants) | 50 | 49
mm | 6.44 (2.83) | 6.14 (2.35)

ADVERSE EVENTS:
Arm/Group | Regular Ibuprofen Dosing | PRN Ibuprofen Dosing
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 2/50 | 2/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regular Ibuprofen Dosing (N=50) | PRN Ibuprofen Dosing (N=49)
nausea and abdominal pain (Gastrointestinal disorders) | 2 (6) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes